CLINICAL TRIAL: NCT01210014
Title: Zinc Sulphate in Treatment of Recurrent Aphthous Stomatitis
Brief Title: Systemic Zinc Sulphate in Treatment of Recurrent Aphthous Ulcerations:A Doubleblind, Placebo Controled Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Qazvin university of medical sciences (dental school), Qazvin university of medical sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QUMS320
Record Dates: First submitted 2010-09-02; First posted 2010-09-28 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Aphthous Stomatitis
Keywords: Recurrent aphthous stomatitis; treatment; zinc sulphate
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): Patients with Recurrent aphthous stomatitis
  Interventions: Drug: placebo: one dosage
- B (Active Comparator): Patients with Recurrent aphthous stomatitis
  Interventions: Drug: zinc sulphate 220mg/day in one dosage

INTERVENTIONS:
Drug: zinc sulphate 220mg/day in one dosage — patients with clinical signs and symptoms of RAS , in whom clinical diagnosis was accompanied with low level of zinc serum were selected for the study. Gender, age, medical history, symptoms, types and site, number, size, pain level, intervals, disease duration and form of treatment were recorded for all participants. Patients were randomly divided into two groups . The case group (n=7) received a single dose of zinc sulphate in the form of 220 mg capsules for 1 month ,while starch-containing placebo was administered with the same dosage and period in the control group.
  The clinical data were scored according to the size of lesions were scored subjectively.
  the symptomatology score was obtained using a visual analogue scale(VAS). All participants in both groups were examined up to 5 months in order to assess the effectiveness of the treatment. At the end of fifth month the serum zinc level was tested again.
  Arms: B
Drug: placebo: one dosage — patients with clinical signs and symptoms of RAS , in whom clinical diagnosis was accompanied with low level of zinc serum were selected for the study. Gender, age, medical history, symptoms, types and site, number, size, pain level, intervals, disease duration and form of treatment were recorded for all participants. Patients were randomly divided into two groups . The case group (n=7) received a single dose of zinc sulphate in the form of 220 mg capsules for 1 month ,while starch-containing placebo was administered with the same dosage and period in the control group.
  The clinical data were scored according to the size of lesions were scored subjectively.
  the symptomatology score was obtained using a visual analogue scale(VAS). All participants in both groups were examined up to 5 months in order to assess the effectiveness of the treatment. At the end of fifth month the serum zinc level was tested again.
  Arms: A

SUMMARY:
Recurrent aphthous stomatitis (RAS) is one of the most common of oral mucosa diseases that affects approximately 20% of the general population. Despite the fact that clinical, pathologic and therapeutic feature of the disease has been comprehensively studied, the pathophysiology of aphthous ulcers remains incompletely understood.

Zinc is a potent catalyst of wound healing and zinc deficiency may be a common cause of delayed tissue repair. Use of zinc sulfate in promotion wound healing and preservation of epithelial integrity advocated its possible use in the treatment or prevention of recurrent oral ulcers.

The purpose of the present study was to determine of systemic zinc sulphate in the treatment of recurrent aphthous stomatitis.

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS) is a chronic inflammatory disease of man characterized by painful ulceration recurring with varying frequency. The pathophysiology of aphthous ulcers remains partly understood. The primary disorder appears to be the result of activation of the cell-mediated immune system. Aphthous ulcers may have abnormalities in cell communication and epithelial integrity. The diagnosis of aphthous ulcers is primarily clinical. Aphthous ulcers occur on areas of nonkeratinized mucosa of the mouth particularly the buccal mucosa, the labial mucosa, the floor of the mouth, the ventral surface of the tongue, and the soft palate. The treatment of recurrent aphthous stomatitis (RAS) still remains unclear and is based mainly on experimental data. The purpose of therapy include the management of pain and functional injury by suppressing inflammatory responses, in addition to reducing the frequency of recurrences or keeping away from the onset of new ulcers .Zinc has been identified as an important factor in repair of tissue.After considerable searching zinc was recognized as the beneficial impurity and a effective factor in healing .The goal of this study is to present the efficiency of dietary zinc supplements in the rate of Recurrent aphthous stomatitis healing.

ELIGIBILITY:
Inclusion Criteria:

1. A history of Recurrent aphthous stomatitis
2. Patients who had symptoms such as burning sensation, pain
3. Patients not on any immunosuppressive or immunomodulatory treatment .
4. Patients of both sexes over 10 years with recurrent aphthous stomatitis
5. Patients who gave written informed consent
6. Patients who were willing for evaluation after therapy and every 1 month up to 5months

Exclusion Criteria:

1. Participants demonstrating drug consumption in the 7 past months
2. pregnancy or lactation
3. Any kind of localized or systemic disease, especially ulcerative colitis , chorn disease and Bechet's syndrome
4. Smokers
5. patients receiving immunosuppressive treatments or any kind of systemic or local drugs especially systemic antibiotics (in past 2 weeks ) and oral antihistamines( in past month ) were either eliminated or asked to discontinue their treatment for a minimum of one month before entering the investigation.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
improvment of Recurrent Aphthous Ulcerations | 5 months
  To assess the improvment of Recurrent Aphthous Ulceration according to Vissual Analoge Scale

SECONDARY OUTCOMES:
Relief sign &symptom | 5 months
relief clinical features | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Kataun Borhanmojabi, DDS,MSC, Study Chair — QUMS; Touba Karagah, DDS, Principal Investigator — QUMS; Reza Mortazavi, PHD, Study Director — QUMS; Samira Ganbarzade, DDS, Principal Investigator — QUMS
Locations (1):
- Qazvin university of medical sciences, Qazvin, Qazvin Province, Iran